CLINICAL TRIAL: NCT02020486
Title: A Multiple Dose Pharmacokinetic Study of Perampanel in Korean Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2007-K082-047
Record Dates: First submitted 2013-12-04; First posted 2013-12-25 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Healthy
MeSH Terms: interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Experimental
  Interventions: Drug: Perampanel
- Group B (Experimental): Days 1-14: Multiple oral dose of 2 mg perampanel (one 2 mg tablet) Days 15-28: Multiple oral dose of 4 mg perampanel (two 2 mg tablets) Days 29-42: Multiple oral dose of 6 mg perampanel (three 2 mg tablets)
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — 2 mg up to 4 mg
  Arms: Group A
Drug: Perampanel — 2 mg up to 6 mg
  Arms: Group B

SUMMARY:
This study will consist of 2 phases: Pretreatment Phase and Treatment Phase. The Pretreatment Phase will have 2 time points: Screening and Baseline. Subjects will be admitted to the clinical study ward the day before starting the study drug administration (Day -1) for PK and safety assessments during Treatment Phase, and discharged at Day 33 (group A) and Day 47 (group B). Post-test will be done at Day 37 (+/-1), Day 42 (+3) (group A) and Day 51 (+/-1), Day 56 (+3) (group B). Study medication will be administered with 240 mL of room temperature water

ELIGIBILITY:
Inclusion Criteria

Subjects who meet all of the following criteria will be included in the study:

1. Korean healthy adult male volunteers
2. Non-smoking, male subjects aged at least 19 years and no more than 55 years old at the time of informed consent
3. Body Mass Index (BMI) of greater than 18 and less than or equal to 30 kg/m2 at Screening. Note: BMI (kg/m2) = body weight (kg)/[height (m) x height (m)]
4. Male subjects must have had a successful vasectomy (confirmed azoospermia) or they and their female partners are not of childbearing potential or practicing highly effective contraception throughout the study period and for 30 days after study drug discontinuation. No sperm donation is allowed during the study period and for 30 days after study drug discontinuation
5. Provide written informed consent
6. Willing and able to comply with all aspects of the protocol

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from participation in the study:

1. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
2. Evidence of disease that may influence the outcome of the study within 4 weeks prior to dosing; e.g., psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or subjects who have a congenital abnormality in metabolism
3. Any history of gastrointestinal surgery that may affect PK profiles of perampanel, e.g., hepatectomy, nephrotomy, digestive organ resection at Screening and Baseline
4. Evidence of clinically significant organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory determinations. Subjects whose liver enzyme values are outside of the acceptable normal limits will be excluded
5. A prolonged QT/QTc interval (QTc greater than 450 ms) demonstrated on ECG at Screening or Baseline
6. Any suicidal ideation with intent with or without a plan at Screening or within 6 months of Screening
7. Any lifetime suicidal behavior
8. Known history of clinically significant drug allergy at Screening and Baseline
9. Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening and Baseline
10. Known to be human immunodeficiency virus (HIV) positive at Screening
11. Active viral hepatitis (A, B or C) as demonstrated by positive serology at Screening
12. History of drug or alcohol dependency or abuse within the 2 years prior to Screening, or those who have a positive urine drug test or breath (or urine) alcohol test at Screening or Baseline
13. Intake of caffeinated beverages or food within 72 hours prior to dosing
14. Intake of nutritional supplements, juice, and herbal preparations or other foods or beverages that may affect CYP (e.g., alcohol, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice, vegetables from the mustard green family [e.g., kale, broccoli, watercress, collard greens, kohlrabi, brussel sprouts, mustard], and charbroiled meats) within 1 week prior to dosing
15. Intake of herbal preparations containing St. John's Wort within 4 weeks prior to dosing
16. Use of prescription drugs within 4 weeks prior to dosing
17. Intake of over-the-counter (OTC) medications within 2 weeks prior to dosing
18. Currently enrolled in another clinical trial or used any investigational drug or device within 30 days or 5x the half-life, whichever is longer preceding informed consent
19. Receipt of blood products within 4 weeks, or donation of blood within 8 weeks, or donation of plasma within one week of dosing
20. Engagement in strenuous exercise within 2 weeks prior to check-in (e.g., marathon runners, weight lifters, etc.)

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of perampanel in Korean healthy male subjects | Approximately 56 days
  PK analysis will be performed on PK Analysis Set using plasma concentrations of perampanel. Plasma concentrations will be tabulated by nominal sampling time and summarized using summary statistics.

SECONDARY OUTCOMES:
Safety and tolerability of perampanel | Approximately 56 days
  Safety will be assessed by monitoring and recording all adverse events (AEs) and serious adverse events (SAEs), regular monitoring of hematology, blood chemistry and urine values, regular measurement of vital signs, weight, physical examinations and electrocardiograms (ECGs).

CONTACTS AND LOCATIONS:
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea